CLINICAL TRIAL: NCT02579980
Title: Development of Quantitative Imaging Biomarkers for Evaluating Sarcoma Patients
Brief Title: Quantitative Imaging Biomarkers for Sarcoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Lawrence Schwartz, James Picker Professor and Chairman Department of Radiology, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AAAO9603; U54CA168512 (NIH)
Record Dates: First submitted 2015-10-15; First posted 2015-10-20 (Estimated); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Sarcoma
Keywords: Dynamic Contrast Enhanced MRI; Diffusion Weighted MRI; Magnetic Resonance Imaging (MRI)
MeSH Terms: conditions — Sarcoma | interventions — delta 24-sterol reductase; Surgical Procedures, Operative; Transurethral Resection of Bladder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DCE and DWI MRI group (Experimental): Patients will undergo a baseline MR exam at enrollment within 4 weeks prior to scheduled surgery, which will include DW-MRI and DCE-MRI prior to surgery and tumor tissue collection.
  Interventions: Procedure: DCE and DWI MRI; Procedure: Surgery

INTERVENTIONS:
Procedure: DCE and DWI MRI — Dynamic Contrast Enhanced MRI (DCE-MRI) and Diffusion Weighted MRI (DW-MRI): DW-MRI is a technique for quantifying the increase in water diffusion caused by cellular necrosis or apoptosis in tumors within days of therapy. DCE-MRI is frequently used in preclinical and early clinical trial assessment of anti-angiogenic and vascular disrupting compounds, also within hours of therapeutic intervention.
Procedure: Surgery — Standard of care procedure for sarcoma patients
  Other Names: Tumor resection

SUMMARY:
Unless a cancer quickly gets smaller with radiation or chemotherapy, the investigators cannot tell if the treatment is working or not. In this research program, two techniques using magnetic resonance imaging (MRI) scanning will be tested in people who have sarcomas, which are rare cancers starting in muscle, tendons, and bones. These particular MRI tests are called dynamic contrast enhanced MRI and diffusion weighted MRI. These MRI scans allow visualization of how sarcomas are different from the normal organs of the body. These MRI tests will tell us the location of sarcoma and its proximity to other structures, as well as correlation of imaging with pathological characteristics after surgery

DETAILED DESCRIPTION:
Dynamic Contrast Enhanced MRI (DCE-MRI) and Diffusion Weighted MRI (DW-MRI) are imaging approaches that are being utilized in preclinical evaluation as well as clinical trials. DW-MRI is a technique for quantifying the increase in water diffusion caused by cellular necrosis or apoptosis in tumors within days of therapy. DCE-MRI is frequently used in preclinical and early clinical trial assessment of anti-angiogenic and vascular disrupting compounds, also within hours of therapeutic intervention. Evidence of drug efficacy and dose-dependent response has been demonstrated with certain angiogenesis inhibitors. It may also provide useful information for identifying early disease progression, independent of the treatment modality. While these approaches provide additional functional information, they have yet to be validated in sarcoma patients. This study seeks to develop a standardized protocol for performing DCE-MRI and DW-MRI and implement this in a clinical trial of patients with sarcomas who will have surgical resection as part of their standard care. This will allow the accuracy of in vivo MRI measurements to be directly compared to histology as ground truth. The study will also determine the reproducibility of these techniques using repeat baseline imaging as well as evaluate the quantitative changes in these parameters before and after therapy and correlate with histopathology. The collaboration between Columbia University and the University of Utah for this project will allow the existing quantitative MRI approaches to be expanded to a multi-center setting, and will establish a paradigm infrastructure for future expansion to larger scale multi-center therapeutic trials in sarcoma.

ELIGIBILITY:
Inclusion Criteria:

* New diagnosis of de novo sarcoma of all histologies (including soft tissue sarcoma, osteosarcoma, Ewing sarcoma, and chondrosarcoma) confirmed by biopsy
* Scheduled to be treated with surgical resection at the sarcoma or cancer center of participating sites
* Availability of the patient's medical information
* Provide written informed consent for the study
* Eighteen years of age or older
* Ability to remain motionless in MRI scanner for approximately 40 minutes

Exclusion Criteria:

* Patients with contra-indications for contrast enhanced MR exam, including:

  * Cardiac pacemaker or pacemaker wiring in situ
  * Cerebral clips or metal artificial cardiac valves
  * Ossicle prosthesis
  * Conditions that could produce a dangerous situation in the presence of a strong magnetic field: line metallic implants, shrapnel, inability to lie still, and conditions that can worsen inside confined spaces (severe claustrophobia, psychosis)
  * Acute or chronic severe renal disease as determined by glomerular filtration rate (GFR) < 30 ml/min/1.73m2
  * Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Correlation coefficient of Ktrans (DCE MR parameter) and Apparent Diffusion Coefficient (ADC) (DWI MR parameter) with microvessel density obtained from histopathology. | through study completion, an average of 4 weeks
  The primary endpoint of this study is to evaluate the correlation of the estimated in vivo Dynamic Contrast Enhanced and Diffusion weighted MRI parameters with ex vivo histopathologic measurements obtained from tumor tissue. Correlation coefficient (range: -1 to 1).

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence H Schwartz, MD, Principal Investigator — James Picker Professor and Chairman Department of Radiology
Locations (2):
- United States (2):
  - Columbia University Medical Center, New York, New York
  - Huntsman Cancer Institute, University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jacobs MA, Herskovits EH, Kim HS. Uterine fibroids: diffusion-weighted MR imaging for monitoring therapy with focused ultrasound surgery--preliminary study. Radiology. 2005 Jul;236(1):196-203. doi: 10.1148/radiol.2361040312. PMID 15987974
- [Background] Castillo M, Arbelaez A, Smith JK, Fisher LL. Diffusion-weighted MR imaging offers no advantage over routine noncontrast MR imaging in the detection of vertebral metastases. AJNR Am J Neuroradiol. 2000 May;21(5):948-53. PMID 10815675
- [Background] Chenevert TL, Meyer CR, Moffat BA, Rehemtulla A, Mukherji SK, Gebarski SS, Quint DJ, Robertson PL, Lawrence TS, Junck L, Taylor JM, Johnson TD, Dong Q, Muraszko KM, Brunberg JA, Ross BD. Diffusion MRI: a new strategy for assessment of cancer therapeutic efficacy. Mol Imaging. 2002 Oct;1(4):336-43. doi: 10.1162/15353500200221482. PMID 12926229
- [Background] Ei Khouli RH, Jacobs MA, Mezban SD, Huang P, Kamel IR, Macura KJ, Bluemke DA. Diffusion-weighted imaging improves the diagnostic accuracy of conventional 3.0-T breast MR imaging. Radiology. 2010 Jul;256(1):64-73. doi: 10.1148/radiol.10091367. PMID 20574085
- [Background] Herneth AM, Friedrich K, Weidekamm C, Schibany N, Krestan C, Czerny C, Kainberger F. Diffusion weighted imaging of bone marrow pathologies. Eur J Radiol. 2005 Jul;55(1):74-83. doi: 10.1016/j.ejrad.2005.03.031. PMID 15921871
- [Background] Jacobs MA, Ouwerkerk R, Kamel I, Bottomley PA, Bluemke DA, Kim HS. Proton, diffusion-weighted imaging, and sodium (23Na) MRI of uterine leiomyomata after MR-guided high-intensity focused ultrasound: a preliminary study. J Magn Reson Imaging. 2009 Mar;29(3):649-56. doi: 10.1002/jmri.21677. PMID 19243047
- [Background] Jin G, An N, Jacobs MA, Li K. The role of parallel diffusion-weighted imaging and apparent diffusion coefficient (ADC) map values for evaluating breast lesions: preliminary results. Acad Radiol. 2010 Apr;17(4):456-63. doi: 10.1016/j.acra.2009.12.004. PMID 20207316
- [Background] Mintorovitch J, Moseley ME, Chileuitt L, Shimizu H, Cohen Y, Weinstein PR. Comparison of diffusion- and T2-weighted MRI for the early detection of cerebral ischemia and reperfusion in rats. Magn Reson Med. 1991 Mar;18(1):39-50. doi: 10.1002/mrm.1910180106. PMID 2062240
- [Background] Moseley ME, Kucharczyk J, Mintorovitch J, Cohen Y, Kurhanewicz J, Derugin N, Asgari H, Norman D. Diffusion-weighted MR imaging of acute stroke: correlation with T2-weighted and magnetic susceptibility-enhanced MR imaging in cats. AJNR Am J Neuroradiol. 1990 May;11(3):423-9. PMID 2161612
- [Background] Babsky AM, Topper S, Zhang H, Gao Y, James JR, Hekmatyar SK, Bansal N. Evaluation of extra- and intracellular apparent diffusion coefficient of sodium in rat skeletal muscle: effects of prolonged ischemia. Magn Reson Med. 2008 Mar;59(3):485-91. doi: 10.1002/mrm.21568. PMID 18306401
- [Background] Le Bihan D, Breton E, Lallemand D, Aubin ML, Vignaud J, Laval-Jeantet M. Separation of diffusion and perfusion in intravoxel incoherent motion MR imaging. Radiology. 1988 Aug;168(2):497-505. doi: 10.1148/radiology.168.2.3393671.
- [Background] Le Bihan D, Breton E, Lallemand D, Grenier P, Cabanis E, Laval-Jeantet M. MR imaging of intravoxel incoherent motions: application to diffusion and perfusion in neurologic disorders. Radiology. 1986 Nov;161(2):401-7. doi: 10.1148/radiology.161.2.3763909.
- [Background] Szafer A, Zhong J, Gore JC. Theoretical model for water diffusion in tissues. Magn Reson Med. 1995 May;33(5):697-712. doi: 10.1002/mrm.1910330516. PMID 7596275
- [Background] Knight RA, Ordidge RJ, Helpern JA, Chopp M, Rodolosi LC, Peck D. Temporal evolution of ischemic damage in rat brain measured by proton nuclear magnetic resonance imaging. Stroke. 1991 Jun;22(6):802-8. doi: 10.1161/01.str.22.6.802. PMID 2057981
- [Background] Jacobs MA, Ouwerkerk R, Wolff AC, Stearns V, Bottomley PA, Barker PB, Argani P, Khouri N, Davidson NE, Bhujwalla ZM, Bluemke DA. Multiparametric and multinuclear magnetic resonance imaging of human breast cancer: current applications. Technol Cancer Res Treat. 2004 Dec;3(6):543-50. doi: 10.1177/153303460400300603. PMID 15560711
- [Background] Kamel IR, Bluemke DA, Eng J, Liapi E, Messersmith W, Reyes DK, Geschwind JF. The role of functional MR imaging in the assessment of tumor response after chemoembolization in patients with hepatocellular carcinoma. J Vasc Interv Radiol. 2006 Mar;17(3):505-12. doi: 10.1097/01.RVI.0000200052.02183.92. PMID 16567675
- [Background] Chenevert TL, Stegman LD, Taylor JM, Robertson PL, Greenberg HS, Rehemtulla A, Ross BD. Diffusion magnetic resonance imaging: an early surrogate marker of therapeutic efficacy in brain tumors. J Natl Cancer Inst. 2000 Dec 20;92(24):2029-36. doi: 10.1093/jnci/92.24.2029. PMID 11121466
- [Background] Hosseinzadeh K, Schwarz SD. Endorectal diffusion-weighted imaging in prostate cancer to differentiate malignant and benign peripheral zone tissue. J Magn Reson Imaging. 2004 Oct;20(4):654-61. doi: 10.1002/jmri.20159. PMID 15390142
- [Background] Brunberg JA, Chenevert TL, McKeever PE, Ross DA, Junck LR, Muraszko KM, Dauser R, Pipe JG, Betley AT. In vivo MR determination of water diffusion coefficients and diffusion anisotropy: correlation with structural alteration in gliomas of the cerebral hemispheres. AJNR Am J Neuroradiol. 1995 Feb;16(2):361-71. PMID 7726086
- [Background] Herneth AM, Philipp MO, Naude J, Funovics M, Beichel RR, Bammer R, Imhof H. Vertebral metastases: assessment with apparent diffusion coefficient. Radiology. 2002 Dec;225(3):889-94. doi: 10.1148/radiol.2253011707. PMID 12461275
- [Background] Hylton N. Dynamic contrast-enhanced magnetic resonance imaging as an imaging biomarker. J Clin Oncol. 2006 Jul 10;24(20):3293-8. doi: 10.1200/JCO.2006.06.8080. PMID 16829653
- [Background] Miller JC, Pien HH, Sahani D, Sorensen AG, Thrall JH. Imaging angiogenesis: applications and potential for drug development. J Natl Cancer Inst. 2005 Feb 2;97(3):172-87. doi: 10.1093/jnci/dji023. PMID 15687360
- [Background] Padhani AR, Leach MO. Antivascular cancer treatments: functional assessments by dynamic contrast-enhanced magnetic resonance imaging. Abdom Imaging. 2005 May-Jun;30(3):324-41. doi: 10.1007/s00261-004-0265-5. PMID 15688112
- [Background] Rehman S, Jayson GC. Molecular imaging of antiangiogenic agents. Oncologist. 2005 Feb;10(2):92-103. doi: 10.1634/theoncologist.10-2-92. PMID 15709211
- [Background] Devries AF, Griebel J, Kremser C, Judmaier W, Gneiting T, Kreczy A, Ofner D, Pfeiffer KP, Brix G, Lukas P. Tumor microcirculation evaluated by dynamic magnetic resonance imaging predicts therapy outcome for primary rectal carcinoma. Cancer Res. 2001 Mar 15;61(6):2513-6. PMID 11289123
- [Background] Evelhoch J, Garwood M, Vigneron D, Knopp M, Sullivan D, Menkens A, Clarke L, Liu G. Expanding the use of magnetic resonance in the assessment of tumor response to therapy: workshop report. Cancer Res. 2005 Aug 15;65(16):7041-4. doi: 10.1158/0008-5472.CAN-05-0674. PMID 16103049
- [Background] Evelhoch JL, LoRusso PM, He Z, DelProposto Z, Polin L, Corbett TH, Langmuir P, Wheeler C, Stone A, Leadbetter J, Ryan AJ, Blakey DC, Waterton JC. Magnetic resonance imaging measurements of the response of murine and human tumors to the vascular-targeting agent ZD6126. Clin Cancer Res. 2004 Jun 1;10(11):3650-7. doi: 10.1158/1078-0432.CCR-03-0417. PMID 15173071
- [Background] Hoskin PJ, Saunders MI, Goodchild K, Powell ME, Taylor NJ, Baddeley H. Dynamic contrast enhanced magnetic resonance scanning as a predictor of response to accelerated radiotherapy for advanced head and neck cancer. Br J Radiol. 1999 Nov;72(863):1093-8. doi: 10.1259/bjr.72.863.10700827.
- [Background] Kawai A, Sugihara S, Kunisada T, Uchida Y, Inoue H. Imaging assessment of the response of bone tumors to preoperative chemotherapy. Clin Orthop Relat Res. 1997 Apr;(337):216-25. doi: 10.1097/00003086-199704000-00024. PMID 9137193
- [Background] Vanel D, Lacombe MJ, Couanet D, Kalifa C, Spielmann M, Genin J. Musculoskeletal tumors: follow-up with MR imaging after treatment with surgery and radiation therapy. Radiology. 1987 Jul;164(1):243-5. doi: 10.1148/radiology.164.1.3588913.
- [Background] Vanel D, Shapeero LG, Tardivon A, Western A, Guinebretiere JM. Dynamic contrast-enhanced MRI with subtraction of aggressive soft tissue tumors after resection. Skeletal Radiol. 1998 Sep;27(9):505-10. doi: 10.1007/s002560050428. PMID 9809880
- [Background] Uhl M, Saueressig U, van Buiren M, Kontny U, Niemeyer C, Kohler G, Ilyasov K, Langer M. Osteosarcoma: preliminary results of in vivo assessment of tumor necrosis after chemotherapy with diffusion- and perfusion-weighted magnetic resonance imaging. Invest Radiol. 2006 Aug;41(8):618-23. doi: 10.1097/01.rli.0000225398.17315.68. PMID 16829744
- [Background] Bartolozzi C, Lencioni R, Caramella D, Mazzeo S, Ciancia EM. Treatment of hepatocellular carcinoma with percutaneous ethanol injection: evaluation with contrast-enhanced MR imaging. AJR Am J Roentgenol. 1994 Apr;162(4):827-31. doi: 10.2214/ajr.162.4.8141000.
- [Background] Castrucci M, Sironi S, De Cobelli F, Salvioni M, Del Maschio A. Plain and gadolinium-DTPA-enhanced MR imaging of hepatocellular carcinoma treated with transarterial chemoembolization. Abdom Imaging. 1996 Nov-Dec;21(6):488-94. doi: 10.1007/s002619900110. PMID 8875869
- [Background] Murakami T, Nakamura H, Hori S, Tomoda K, Mitani T, Nakanishi K, Hashimoto T, Tsuda K, Kozuka T, Monden M, et al. Detection of viable tumor cells in hepatocellular carcinoma following transcatheter arterial chemoembolization with iodized oil. Pathologic correlation with dynamic turbo-FLASH MR imaging with Gd-DTPA. Acta Radiol. 1993 Jul;34(4):399-403. PMID 8391291
- [Background] Feydy A, Anract P, Tomeno B, Chevrot A, Drape JL. Assessment of vascular invasion by musculoskeletal tumors of the limbs: use of contrast-enhanced MR angiography. Radiology. 2006 Feb;238(2):611-21. doi: 10.1148/radiol.2382041725. PMID 16436820
- [Background] Tofts PS, Brix G, Buckley DL, Evelhoch JL, Henderson E, Knopp MV, Larsson HB, Lee TY, Mayr NA, Parker GJ, Port RE, Taylor J, Weisskoff RM. Estimating kinetic parameters from dynamic contrast-enhanced T(1)-weighted MRI of a diffusable tracer: standardized quantities and symbols. J Magn Reson Imaging. 1999 Sep;10(3):223-32. doi: 10.1002/(sici)1522-2586(199909)10:33.0.co;2-s. PMID 10508281
- [Background] Marcus CD, Ladam-Marcus V, Cucu C, Bouche O, Lucas L, Hoeffel C. Imaging techniques to evaluate the response to treatment in oncology: current standards and perspectives. Crit Rev Oncol Hematol. 2009 Dec;72(3):217-38. doi: 10.1016/j.critrevonc.2008.07.012. Epub 2008 Aug 29. PMID 18760935